CLINICAL TRIAL: NCT06745206
Title: Recombinant Human Brain Natriuretic Peptide for the Recovery Stage of Septic Shock: An Interventional Pilot Study
Brief Title: Recombinant Human Brain Natriuretic Peptide for the Recovery Stage of Septic Shock
Acronym: rh-BNP-RSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Collaborators: Tibet Kangzhe Pharmaceutical Development Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Lingai Pan, associate chief physician, Sichuan Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-653-1
Record Dates: First submitted 2024-12-09; First posted 2024-12-20 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Sepsis-induced Cardiomyopathy; the Recovery Phase of Septic Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rh-BNP arm (Experimental): rh-BNP is reconstituted to a concentration of 10 μg/mL and administered as an initial intravenous bolus of 2 μg/kg over 15 minutes, followed by a continuous infusion at a rate of 0.01 μg/kg/min. Patients should receive at least the first 500μg dose infusion, with a recommended duration of 72 hours. The specific timing of discontinuation will be determined by the attending physician.
  Interventions: Drug: Lyophilized Recombinant Human Brain Natriuretic Peptide

INTERVENTIONS:
Drug: Lyophilized Recombinant Human Brain Natriuretic Peptide — rh-BNP is reconstituted to a concentration of 10 μg/mL and administered as an initial intravenous bolus of 2 μg/kg over 15 minutes, followed by a continuous infusion at a rate of 0.01 μg/kg/min. Patients should receive at least the first 500μg dose infusion, with a recommended duration of 72 hours. The specific timing of discontinuation will be determined by the attending physician. Prior to rh-BNP administration, measure: PiCCO indices, hemodynamic parameters, venous return, tissue perfusion, echocardiographic parameters, ultrasound indices, 2-hour averaged urine output and fluid balance. Repeat all above-mentioned measurements at 30 minutes post-initiation.
  Other Names: S20050033

SUMMARY:
As infection control improves and circulation stabilizes, treatment de-escalation of septic shock begins, accompanied by fluid redistribution from interstitial spaces to the vasculature, increasing cardiac volume load. Synthetic recombinant human BNP (rh-BNP) plays a role in inducing vasodilation, particularly in the venous system, alleviating cardiac congestion, and enhancing natriuresis and diuresis. Thus the investigators designed a single-center, prospective physiological study to evaluate the efficacy of standard rh-BNP infusion in reducing venous return and enhancing fluid removal, with a secondary objective of assessing the maintenance of perfusion pressure and tissue perfusion.

ELIGIBILITY:
Inclusion criteria:

1. Age >18 years.
2. Septic shock in recovery phase with decreasing vasopressor requirements, which is defined as:

   1. Fulfilling the Sepsis-3 definition of septic shock at initial stage.
   2. Hemodynamic stability achieved after adequate initial resuscitation and individualized hemodynamic optimization.
   3. Controlled infection source with 48-hour trend of improving temperature, white blood cell count, and procalcitonin.
   4. 48-hour trend of decreasing vasopressor requirements and transition to negative fluid balance.
   5. Adequate perfusion with warm extremities, and capillary refill time <3 seconds.
3. Ongoing pulse index continuous cardiac output (PiCCO) hemodynamic monitoring and sinus rhythm.
4. Volume indicators above the lower limit of normal range, with global end-diastolic volume index (GEDI) >680 mL/m2 and central venous pressure (CVP) >8 mmHg.
5. Signs of cardiac dysfunction: BNP>200[10] or NT-proBNP >900 pg/ml[6] or reduced ejection fraction (LVEF) < 50%.
6. No bolus dose of diuretics had been administered in the previous 6 hours.
7. Informed consent obtained from patient/legal representative.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Arrhythmia.
3. Advanced renal dysfunction (Acute Kidney Injury [AKI] stage 3 or Chronic Kidney Disease [CKD] stage 3b or higher) based on Kidney Disease: Improving Global Outcomes (KDIGO) criteria.
4. Inadequate ultrasound window preventing acquisition of diagnostic-quality images.
5. Trauma or neurological diseases (including intracerebral hemorrhage and cerebral infarction).
6. Pre-existing severe heart failure (New York Heart Association [NYHA] class III-IV) or acute myocardial infarction within the past 30 days.
7. Concurrent enrollment in interventional trials that could confound study outcomes.

Criteria for withdrawing from the study:

1. Withdrawal of the informed consent.
2. Severe hemodynamic deterioration necessitating the discontinuation of all vasodilatory medications.
3. Treating clinician's decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The pressure gradient of venous return | From baseline to 30 minutes after rh-BNP initiation.
  Pmsf - CVP

SECONDARY OUTCOMES:
Perfusion pressure | From baseline to 30 minutes, 24 hours, 48 hours and 72 hours after rh-BNP initiation.
  Absolute and relative changes in perfusion pressure (MAP - CVP)
CVP | From baseline to 30 minutes, 24 hours, 48 hours and 72 hours after rh-BNP initiation.
  Absolute and relative changes in CVP
GEDI and global and left-ventricular preload (LVEDV) | From baseline to 30 minutes, 24 hours, 48 hours and 72 hours after rh-BNP initiation.
  Absolute and relative changes in GEDI and global and left-ventricular preload (LVEDV)
Renal microvascular resistance | From baseline to 30 minutes, 24 hours, 48 hours and 72 hours after rh-BNP initiation.
  Absolute and relative changes in renal microvascular resistance
Lactate clearance | From baseline to 30 minutes, 24 hours, 48 hours and 72 hours after rh-BNP initiation.
  Absolute and relative changes in lactate clearance
Duration of invasive mechanical ventilation | From baseline to 30 minutes, 24 hours, 48 hours and 72 hours after rh-BNP initiation.
  Duration of invasive mechanical ventilation
ICU lengths of stay | From baseline to 30 minutes, 24 hours, 48 hours and 72 hours after rh-BNP initiation.
  ICU lengths of stay

OTHER OUTCOMES:
Safety outcome | From baseline to 30 minutes, 24 hours, 48 hours and 72 hours after rh-BNP initiation.
  The safety outcome was hemodynamic instability, defined as a sustained (≥15 minutes) decrease in systolic blood pressure ≥ 10 mmHg or MAP ≥ 5 mmHg compared with baseline, or a requirement for ≥ 0.1 µg/kg/min increase in norepinephrine to maintain MAP ≥ 65 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Lingai Pan, MD, Principal Investigator — Sichuan Academy of Medical Sciences and Sichuan Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No